CLINICAL TRIAL: NCT03190031
Title: Respiratory Muscle Training in Patients With Cystic Fibrosis
Brief Title: Respiratory Muscle Training in CF Patients
Acronym: MUCOMUREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01652-49
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis; Respiratory Muscles
Keywords: training; exercise; quality of life
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: The patients will be randomized in 2 different groups, one being involved in an endurance respiratory muscle training program, the other being involved in resistance inspiratory muscle training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endurance respiratory muscle training (Experimental): The intervention consists in performing isocapnic hyperpnea at 70-80% of maximal voluntary ventilation for 20 min, 5 times a week, for 8 weeks
  Interventions: Other: Endurance respiratory muscle training
- Resistance inspiratory muscle training (Active Comparator): The intervention consists in performing inspiratory resistive breathing at 70-80% of maximal inspiratory pressure for 20 min, 5 times a week, for 8 weeks
  Interventions: Other: Resistance inspiratory muscle training

INTERVENTIONS:
Other: Endurance respiratory muscle training — Training program of the respiratory muscles in endurance by using sustained isocapnic hyperpnea
  Arms: Endurance respiratory muscle training
Other: Resistance inspiratory muscle training — Training program of the inspiratory muscles in resistance by using repeated inspiratory maneuvers against a resistance
  Arms: Resistance inspiratory muscle training

SUMMARY:
The present study aims at evaluating the effect of respiratory muscle training in adult patients with cystic fibrosis on lung function, exercise performance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of cystic fibrosis
* Patients in steady state

Exclusion Criteria:

* Patients during exacerbation
* Patients treated by oral corticotherapy (>0.5 mg/kg/j during >7 days) during the past 2 months
* Pregnant patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle endurance | Change from baseline (i.e. T0) measured immediately after the 8 weeks of intervention (T1)
  Total breathing duration (in min) measured during an incremental hyperpnea test

SECONDARY OUTCOMES:
Respiratory muscle strength | Change from baseline (i.e. T0) measured immediately after the 8 weeks of intervention (T1)
  Peak pressure (in mmHg) during maximal inspiratory and expiratory maneuvers
Maximal cycling performance | Change from baseline (i.e. T0) measured immediately after the 8 weeks of intervention (T1)
  Peak maximal power output (in W) during an incremental cycling test
Quality of life of patients after the intervention | Change from baseline (i.e. T0) measured immediately after the 8 weeks of intervention (T1)
  Score obtained during the questionnaire CQF14+

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stanford G, Ryan H, Solis-Moya A. Respiratory muscle training for cystic fibrosis. Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD006112. doi: 10.1002/14651858.CD006112.pub5. PMID 33331663